CLINICAL TRIAL: NCT00954382
Title: Trends in Intellectual Development, and Diverging Verbal and Non-verbal Abilities in the Down Syndrome Phenotype
Brief Title: Trends in Intellectual Development in Down Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Hwu Wuh-Liang, Department of Pediatrics and Medical Genetics, NTUH
Other Study IDs: 200904037R
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Down Syndrome
Keywords: Down syndrome; IQ; mental age; neuropsychological function
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IQ trend: all subjects

SUMMARY:
Previous foreign studies revealed that the IQ in Down syndrome (DS) declines with age, but not any investigation of domestic data in Taiwan was available. Individuals with DS are characterized by limited verbal development, and in this article, authors look into the diverging verbal-nonverbal abilities in the DS phenotype.

DETAILED DESCRIPTION:
The present study investigated this by analysis the test results of development /intelligence scales. To compare initial cross-sectional data with longitudinal follow-up, about 12 people with DS were included.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome with psychological test results

Exclusion Criteria:

* Comorbidity of severe Autism or visual/auditory impairment

Ages: 3 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Down syndrome
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
IQ | 2001-2010

SECONDARY OUTCOMES:
mental age | 2001-2010

CONTACTS AND LOCATIONS:
Overall Officials: Wuh-Liang Hwu, Ph.D., Principal Investigator — NTUH
Locations (1):
- NTUH, Taipei, Taiwan